## THE EFFECT OF NURSING INTERVENTIONS BASED ON CONSERVATION MOTIVATION THEORY ON DRUG ADHERENCE AND HEALTHY LIFESTYLE BEHAVIORS IN PATIENTS WITH HYPERTENSION: A RANDOMIZED CONTROLLED STUDY

NCT05995977

**Document Date: 1 November 2023** 

## Patient information and consent form

Designed for the study titled "The Effect of Nursing Interventions Based on the Theory of Protection Motivation on Medication Adherence and Healthy Lifestyle Behaviors in Hypertensive Patients: A Randomized Controlled Study"

Despite the availability of effective lifestyle changes and drug treatments today, the increasing prevalence of hypertension suggests that people do not understand the seriousness and importance of their diseases and easily ignore the current information given to them. In this context, it is thought that the nursing intervention to be used in our study will adopt effective medication adherence and healthy lifestyle behaviors for the effective management of hypertension. Therefore, I invite you to "Nursing Interventions", which include hypertension education and sending SMS messages. In the study, you are asked to allocate approximately 1 hour of hypertension education and then 12 weeks of SMS messages. Participation in this study is completely voluntary. In order for the study to achieve its purpose, it is expected from you to answer all questions completely, without being under anyone's pressure or suggestion, and sincerely giving the answers that seem most appropriate to you. By reading and approving this form, you agree to participate in the study. However, you also have the right not to participate in the study or to stop the study at any time after participating. The information obtained from this study will be used solely for research purposes and your personal information will be kept confidential; however, your data may be used for publication purposes. If you would like the general/specific results to be shared with you when the study is completed, please let the researcher know.

## ASSISTANT RESEARCHER

Handan ALTUNKAN Karaman Provincial Health Directorate

Telephone: 0536744 3152

Signature:

| ☐ I Want to Participate in the Research |
|-----------------------------------------------|
| □ I Don't Want to Participate in the Research |
| Participant's Name and Surname: |
| Date: |

## **RESPONSIBLE RESEARCHER:**

Doç.Dr. Dilek CİNGİL Necmettin Erbakan University Faculty of Nursing Meram/KONYA Telephone: 0332 3204049